CLINICAL TRIAL: NCT01314092
Title: Phase II Study to Evaluate Efficacy and Safety of ANTG-ASC (Autologous Cultured Adipose-derived Stem Cells) on the Complex Fistula Patients
Brief Title: Clinical Trials of Autologous Cultured Adipose-derived Stem Cells (ANTG-ASC) on Complex Fistula
Acronym: ANTG-ASC-210
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty recruiting subjects.
Sponsor: Anterogen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANTG-ASC-210
Record Dates: First submitted 2011-03-08; First posted 2011-03-14 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2011-03

CONDITIONS: Complex Perianal Fistula
Keywords: crohn's disease; fistula; complex
MeSH Terms: conditions — Crohn Disease; Fistula | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Low dose group
  Interventions: Biological: Autologous cultured adipose derived stem cells(low dose group)
- Group 2 (Experimental): high dose group
  Interventions: Biological: Autologous cultured adipose derived stem cells(high dose group)

INTERVENTIONS:
Biological: Autologous cultured adipose derived stem cells(low dose group) — low dose group: 1x10e7 cells/mL At 6 weeks after first stem cell injection, fistula closing was assessed. If it is not completely closed, second injection would be applied in 2 weeks. Additional dosage would be doubled to first dosage.
  Other Names: mesenchymal stem cell, ANTG-ASC, adipose derived stem cell; Group1: low dose group
  Arms: Group 1
Biological: Autologous cultured adipose derived stem cells(high dose group) — high dose group: 2x10e7 cells/mL At 6 weeks after first stem cell injection, fistula closing was assessed. If it is not completely closed, second injection would be applied in 2 weeks. Additional dosage would be doubled to first dosage.
  Other Names: mesenchymal stem cell, ANTG-ASC, adipose derived stem cell; Group2: high dose group
  Arms: Group 2

SUMMARY:
Mesenchymal stem cells derived from adipose tissue are pluripotent to differentiate into myocytes, adipocytes or others. They have an immunosuppressive activity. Complex perianal fistula is difficult to cure and easy to relapse. Autologous adipose stem cells have shown efficacy and safety on Crohn's fistula in phase 1 study. Based on these results, the investigators would apply autologous adipose stem cells on complex perianal fistula to evaluate their efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* a patient who has complex perianal fistula
* a patient who is negative in pregnancy test
* a patient who has submitted a written consent

Exclusion Criteria:

* a patient who has participated in other clinical studies within 30 days before this clinical trial or has not passed 5 fold period of a half-life of other investigational drugs.
* a patient who has a history of variant Creutzfeldt Jacobs disease or related diseases
* a patient who is allergic to anesthetics, bovine derived proteins or a fibrin glue
* a patient who has an autoimmune disease
* a patient who has infectious diseases such as hepatitis B virus (HBV), hepatitis C virus (HCV) or human immunodeficiency virus (HIV)
* a patient who has sepsis or active tuberculosis
* a patient who is pregnant or breast feeding
* a patient who has inflammatory Bowel disease
* over 2cm in diameter of fistula

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with complete closure of fistula (week 8) | 8 weeks
  Proportion of patients with completely closed fistula (week 8)

SECONDARY OUTCOMES:
Grade of investigator's satisfaction | 8 weeks
  Grade of investigator's satisfaction (8 weeks after final dose)
  1. very satisfaction
  2. satisfaction
  3. somewhat satisfaction
  4. unsatisfaction
  5. very unsatisfaction
Number of patients with closed fistula | 8 weeks
  * proportion of patients with completely closed fistula (every visits)
  * proportion of patients with more than 50 % closed fistula (every visits)
Photo of target fistula | 8 weeks
  Taking picture of target fistula at Day 0 and Week 4, 6, 8
Number of patients with adverse events | 8 weeks
  Number of patients with any kinds of adverse events (Day 0, every visits)

CONTACTS AND LOCATIONS:
Overall Officials: KJ Park, MD, PhD, Principal Investigator — Seoul National University Hospital; DS Kim, Principal Investigator — Daehang Hospital
Locations (6):
- South Korea (6):
  - Soon cheun Hyang university bucheon hospital, Bucheon-si
  - Ewha womwn university mokdong hospital, Seoul
  - DaeHang Hospital, Seoul
  - Samsung seoul Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul Saint Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided